CLINICAL TRIAL: NCT07260643
Title: Valuation of Laser-Assisted (SiLaC®) Technique for the Management of Pilonidal Sinus in Adults: A Prospective Single-Center Cohort at Hospital Universitario La Paz.
Brief Title: SiLaC Laser Technique for Pilonidal Sinus - La Paz Cohort Study.
Acronym: SiLaC-LaPaz
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Luis Asensio Gomez, Consultant, Hospital Universitario La Paz
Other Study IDs: Hospital Universitario La Paz
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Pilonidal Sinus Disorder; Pilonidal Cyst Without Abscess; Pilonidal Sinus; Pilonidal Cysts; Pilonidal Sinus Treatment
Keywords: Pilondal sinus; Pilonidal Cyst; SilaC; laser-assisted closure; minimal invasive surgery; coloproctology; postoperative recovery
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SilaC: Single cohort including all consecutive adult patients operated on using the SiLaC technique between August 2024 and January 2026. Data collected retrospectively and prospectively from clinical records and follow-up interviews
  Interventions: Procedure: SilaC

INTERVENTIONS:
Procedure: SilaC — The SiLaC procedure is a minimally invasive laser technique for the management of chronic pilonidal sinus. It uses a 1470-nm diode laser radial fiber to ablate the sinus tract epithelium after curettage, inducing concentric contraction of the cavity. In this study, patients are observed as part of routine clinical care; the procedure is not assigned or modified by the study protocol.

SUMMARY:
Pilonidal sinus disease (PSD) is a chronic inflammatory condition of the sacrococcygeal region that frequently affects young adults, often causing pain, drainage, and recurrent infection. Traditional surgical approaches such as wide excision or flap techniques may result in prolonged healing times, relevant postoperative pain, and recurrence rates up to 20-30%.

The SiLaC (Sinus Laser-Assisted Closure) technique is a minimally invasive procedure that uses a 1470-nm diode laser fiber to ablate the sinus epithelium and induce concentric contraction of the tract. International studies have reported promising results with faster recovery, minimal wound care, and low morbidity.

This prospective single-center cohort study aims to evaluate the clinical outcomes and perceived recovery time of adult patients treated with the SiLaC® technique at Hospital Universitario La Paz (Madrid, Spain). The main outcome is the total recovery time perceived by patients after surgery. Secondary outcomes include postoperative complications, recurrence rate, pain intensity, need for wound care, and patient satisfaction. Data will be collected from medical records and structured follow-up interviews.

DETAILED DESCRIPTION:
Pilonidal sinus disease (PSD) represents a chronic, recurrent inflammatory disorder of the natal cleft that primarily affects young males. It is associated with risk factors such as obesity, prolonged sitting, and deep gluteal folds. Although not life-threatening, PSD significantly affects quality of life and healthcare resources due to recurrences and delayed wound healing.

Conventional surgical approaches, including excision with secondary healing or flap reconstruction (Limberg, Karydakis, Bascom), often require prolonged recovery and intensive postoperative care. Minimally invasive alternatives have been developed to improve patient recovery and reduce morbidity. Among them, the SiLaC® (Sinus Laser-Assisted Closure) technique employs a radial 1470-nm diode laser fiber to achieve epithelial destruction and tract contraction after curettage. Early evidence suggests favorable outcomes, but robust prospective data remain scarce, especially in Spain.

This study is an ambispective, descriptive, single-center cohort conducted at Hospital Universitario La Paz, Madrid. It includes all adult patients (≥18 years) who undergo SiLaC® surgery for chronic pilonidal sinus between August 2024 and January 2026. Data will be collected retrospectively from electronic health records and prospectively during follow-up visits and structured interviews.

The primary outcome is the total recovery time perceived by the patient (days from surgery to full return to normal activities).

Secondary outcomes include postoperative complications (minor or major), pain intensity (EVA 0-10), wound infection, recurrence within 6 months, patient satisfaction (0-10 scale), and number of wound care visits.

Data will be anonymized and analyzed descriptively using R software (version 4.3.1). Normality will be assessed with the Kolmogorov-Smirnov test; comparisons will use Student's t-test, Mann-Whitney, ANOVA, or Chi-square as appropriate. A significance level of p < 0.05 will be applied.

The study poses no additional risk, as SiLaC® is part of routine surgical practice. Ethical approval will be obtained from the Institutional Ethics Committee (CEIm of Hospital Universitario La Paz / IdiPAZ). Patient confidentiality will be guaranteed under EU Regulation 2016/679 and Spanish Law 3/2018.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Clinical diagnosis of chronic pilonidal sinus disease.
* Undergoing surgery using the SiLaC (Sinus Laser-Assisted Closure) technique.
* Signed informed consent for the use of anonymized clinical data for research purposes.

Exclusion Criteria:

* Patients with inflammatory bowel disease or complex anorectal fistulas.
* Severe immunosuppression (active chemotherapy, high-intensity immunosuppressive therapy, uncontrolled HIV).
* Prior pelvic radiotherapy.
* Missing essential clinical data required for outcome assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with chronic pilonidal sinus disease who undergo laser-assisted closure (SiLaC®) at the Department of General and Digestive Surgery, Coloproctology Section, Hospital Universitario La Paz (Madrid, Spain). Participants will be included consecutively between August 2024 and January 2026, with a minimum follow-up of 6 months after surgery.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Total perceived recovery time | 90 days
  Number of days from surgery to full return to normal activities, as reported by the patient during follow-up interviews

SECONDARY OUTCOMES:
Postoperative complications | 30 days
  Any adverse event (infection, seroma, hematoma, abscess, persistent pain ≥ EVA 4, reintervention).
Pain intensity | 7 days
  Pain intensity measured using the Visual Analog Scale for pain (VAS), a 0-10 scale where 0 indicates 'no pain' and 10 indicates 'worst imaginable pain'. Higher scores reflect worse pain. Pain will be assessed at 24-48 hours and on postoperative day 7
recurrence | 90 days
  Reappearance of drainage, fistulous orifices, or need for a new procedure after initial healing
Need for local wound care | 30 days
  Number of dressing visits at hospital or primary care center

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. The study uses anonymized clinical data stored in institutional repositories at Hospital Universitario La Paz/IdiPAZ. Data access is restricted to the research team in compliance with EU Regulation 2016/679 (GDPR) and Spanish data protection law.